CLINICAL TRIAL: NCT06625177
Title: A Phase 1b, Open-Label Trial to Assess Safety and Exploratory Efficacy of TEV-53408 in Participants With Vitiligo
Brief Title: A Trial to Test the Safety and Efficacy of TEV-53408 in Treating Vitiligo
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV53408-IMM-10209
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TEV-53408 (Experimental): solution administered subcutaneously
  Interventions: Drug: TEV-53408

INTERVENTIONS:
Drug: TEV-53408 — TEV-53408 injection administered subcutaneously

SUMMARY:
The primary objective of the trial is to evaluate the safety of TEV-53408 administered subcutaneously for the treatment of adults with vitiligo.

A secondary objective is to further evaluate the safety of TEV-53408.

The planned study period per participant is 84 weeks including a screening period (up to 4 weeks), a 24-week open-label treatment period, a 16-week washout period, and a 40-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of active or stable vitiligo for at least 3 months.
* The participant has a body mass index (BMI) within the range of 18.5 to 40.0 kg/m2
* A female participant is eligible if she is not pregnant or breastfeeding AND is a woman of nonchildbearing potential OR is a women of childbearing potential using a contraceptive method that is highly effective AND agrees not to donate eggs for the purpose of reproduction for the required period
* A male participant is eligible if he agrees to refrain from donating sperm PLUS remain abstinent from heterosexual intercourse OR use a male condom with a female partner for the required period
* The participant is capable of giving signed, informed consent
* The participant agrees to discontinue all agents and procedures used to treat vitiligo during the treatment period in the trial
* If receiving permitted concomitant medications for any reason other than vitiligo, the participant must be on a stable regimen,
* The participant must agree to avoid prolonged exposure to the sun, must use sunscreen, and must not use tanning booths, sun lamps, or other ultraviolet light sources

NOTE - Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant suffers from vitiligo induced by exposure to chemicals or immunotherapy known to induce vitiligo
* The participant has other autoimmune diseases for which systemic immunotherapy is or may be warranted
* The participant has current or history of malignancy or treatment of malignancy in the last 5 years, excluding fully-treated basal cell carcinoma
* Infectious disease
* The participant has used skin bleaching treatments for past treatment of vitiligo or other pigmented areas
* The participant has a history of melanocyte-keratinocyte transplantation procedure or other surgical treatment for vitiligo. After 2 or more years since last melanocyte-keratinocyte transplantation procedure, the participants may be included in the trial.
* The participant has donated or received any blood or blood products (white blood cells, platelets, etc) within the 60 days prior to screening or has donated blood or blood products on 2 or more occasions within the 6 months prior to IMP administration, or has donated plasma within 7 days before the screening visit, or has planned donations during the trial
* The participant has current or history of alcohol or other substance abuse

NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With at Least One Treatment-Emergent Adverse Event | Up to Week 40
Number of Participants With at Least One Serious Treatment-Emergent Adverse Event | Up to Week 40
Number of Participants With at Least One Protocol-Defined Adverse Event of Special Interest | Up to Week 40
Number of Participants With at Least One Treatment-Related Adverse Event | Up to Week 40
Number of Participants who Discontinued Treatment due to an Adverse Event | Up to Week 40

SECONDARY OUTCOMES:
Number of Participants With at Least One Protocol-Defined Adverse Event of Special Interest | Week 40 to Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D LLC
Locations (13):
- United States (13):
  - Teva Investigational Site 12043, Scottsdale, Arizona
  - Teva Investigational Site 12052, Hot Springs, Arkansas
  - Teva Investigational Site 12044, Fremont, California
  - Teva Investigational Site 12051, Irvine, California
  - Teva Investigational Site 12046, Pasadena, California
  - Teva Investigational Site 12049, Miramar, Florida
  - Teva Investigational Site 12047, Chicago, Illinois
  - Teva Investigational Site 12053, Louisville, Kentucky
  - Teva Investigational Site 12048, Canton, Michigan
  - Teva Investigational Site 12054, Portland, Oregon
  - Teva Investigational Site 12045, Dallas, Texas
  - Teva Investigational Site 12057, Webster, Texas
  - Teva Investigational Site 12055, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.